CLINICAL TRIAL: NCT00120250
Title: Eszopiclone for Sleep Disturbance and Nightmares in Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mark H. Pollack, Grainger Professor and Chairman, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-P-000645
Record Dates: First submitted 2005-07-07; First posted 2005-07-15 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-03

CONDITIONS: Post-Traumatic Stress Disorders
Keywords: PTSD; Sleep disturbance; Eszopiclone; Double-blind; Crossover
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Parasomnias | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eszopiclone (Experimental): Subjects received 3mg eszopiclone nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of placebo, followed by another 1 week washout.
  Interventions: Drug: Eszopiclone
- Placebo (Placebo Comparator): Subjects received placebo nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of 3mg eszopiclone, followed by another 1 week washout.
  Interventions: Drug: Eszopiclone

INTERVENTIONS:
Drug: Eszopiclone — The total study duration is 8 weeks, with subjects receiving 3mg eszopiclone or placebo nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of the alternate condition, followed by another 1 week washout.
  Other Names: Lunesta

SUMMARY:
The purpose of this study is to obtain data investigating the safety and efficacy of eszopiclone for the treatment of post-traumatic stress disorder (PTSD)-related sleep disturbance and the impact of improved sleep with eszopiclone treatment on neuroendocrine correlates of PTSD. The investigators hypothesize that eszopiclone will be significantly more effective than placebo and well tolerated for PTSD-related sleep disturbance, improvement in sleep will be associated with improvement in overall PTSD symptoms, and patients with PTSD-related sleep disturbances will have abnormal levels of stress hormones.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is characterized by three symptom groupings: re-experiencing symptoms including flashbacks, nightmares, and intrusive memories; physiological hyperarousal; and avoidance symptoms. Of the three major categories of symptoms in PTSD listed by the Diagnostic and Statistical Manual of Mental Disorders, sleep-related problems are listed in two of them: difficulty falling asleep is considered an aspect of hyperarousal symptoms, and nightmares are a type of re-experiencing symptom. Both are found commonly in PTSD. Little is known about the relationship of neuroendocrine dysregulation in PTSD and sleep disturbance. It is possible that successful treatment of sleep disturbance in PTSD may alter an abnormal stress hormone pattern. The novel cyclopyrrolone hypnotic eszopiclone thus presents an intriguing opportunity to examine the treatment of sleep disturbances and nightmares in PTSD. This study will determine the safety, efficacy and impact on neuroendocrine parameters of eszopiclone compared to placebo for sleep disturbance and overall PTSD symptoms in individuals with PTSD and reported sleep disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18-64 years of age with a primary diagnosis of PTSD as defined by DSM-IV criteria with associated sleep disturbance

Exclusion Criteria:

* Pregnant women, lactating women, and women of childbearing potential who are not using medically accepted forms of contraception.
* Concurrent use of other psychotropic medications, other than antidepressants at stable dose for at least 4 weeks prior to randomization
* Serious medical illness or instability
* Seizure disorders with the exception of a history of febrile seizures if they occurred during childhood
* Concurrent psychotherapy initiated within one month of randomization or ongoing psychotherapy of any duration directed specifically toward treatment of PTSD and/or sleep disturbance
* Diagnosis of schizophrenia, mental retardation, OCD, organic medical disorders or bipolar disorder, eating disorders in the past 6 months, alcohol or substance abuse in the past 3 months, or dependence within the past 6 months.
* Patients with significant suicidal ideation or who have enacted suicidal behaviors within 6 months prior to intake

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pollack, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Pollack MH, Hoge EA, Worthington JJ, Moshier SJ, Wechsler RS, Brandes M, Simon NM. Eszopiclone for the treatment of posttraumatic stress disorder and associated insomnia: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2011 Jul;72(7):892-7. doi: 10.4088/JCP.09m05607gry. Epub 2011 Feb 22. PMID 21367352
- See also: Official Website for the Center for Anxiety and Traumatic Stress Disorders — http://www.mghanxiety.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Eszopiclone, Then Placebo: The total study duration is 8 weeks, with subjects receiving 3mg eszopiclone nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of placebo, followed by another 1 week washout.
- Placebo, Then Eszopiclone: The total study duration is 8 weeks, with subjects receiving placebo nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of 3mg eszopiclone, followed by another 1 week washout.
Period: Overall Study
Arm/Group | Eszopiclone, Then Placebo | Placebo, Then Eszopiclone
Started | 13 | 14
Completed | 12 | 12
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data are unavailable for the 3 participants that did not complete the study, and therefore, the baseline data will only reflect the information of the 24 completed participants, instead of the 27 that began baseline.
Groups:
- Drug vs Placebo: Eszopiclone : The total study duration is 8 weeks, with subjects receiving 3mg eszopiclone or placebo nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of the alternate condition, followed by another 1 week washout.
Arm/Group | Drug vs Placebo
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.0 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Short PTSD Rating Interview (SPRINT)
Description: The SPRINT is a 8-item, clinician-administered scale assessing core and related symptoms of PTSD. Symptoms are rates on 5 point scales from 0 (not at all) to 4 (very much) where a higher value indicates a worse outcome.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: The total study duration is 8 weeks, with subjects receiving 3mg eszopiclone or placebo nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of the alternate condition, followed by another 1 week washout.
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 16.13 (4.56) | 19.88 (5.47)

2. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The PSQI is a 24-item, patient-administered scale that assess changes in sleep symptomatology. The total PSQI score ranges from 0 to 21 where a higher value indicates a worse sleep symptomatology.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 24 | 24
units on a scale | 8.30 (3.28) | 11.29 (3.86)

3. Secondary Outcome: Sleep Latency
Description: Sleep Latency was derived from a subject-completed daily sleep diary.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 24 | 24
Minutes | 25.83 (17.55) | 55.83 (82.39)

4. Secondary Outcome: Total Sleep Time
Description: Total Sleep Time was derived from a subject-completed daily sleep diary.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 24 | 24
Minutes | 390 (83.46) | 362.38 (67.3)

5. Secondary Outcome: Clinician-Administered PTSD Scale (CAPS)
Description: The CAPS is a highly detailed measure of the presence and severity of the DSM-IV PTSD criteria. The severity score was calculated by adding up the frequency score (scale 0 = "none of the time" to 4 = "most or all of the time") and an intensity score (scale 0 = "none" to 4 = "extreme"), which can then be summed for all 17 symptom questions and/or for the three symptom clusters. Scores range from 0 to 136, where greater than or equal to 80 represents extreme PTSD symptomatology. In this case, the total score for all 17 symptom questions, which is also the sum of the three symptom clusters, is used.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Eszopiclone: The total study duration is 8 weeks, with subjects receiving 3mg eszopiclone nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of placebo, followed by another 1 week washout.
- Placebo: The total study duration is 8 weeks, with subjects receiving placebo nightly for 3 weeks, followed by a 1 week washout period, followed by 3 weeks of 3mg eszopiclone, followed by another 1 week washout.
Arm/Group | Eszopiclone | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 53.92 (17.05) | 67.5 (20.83)

ADVERSE EVENTS:
Arm/Group | Drug vs Placebo
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No